CLINICAL TRIAL: NCT07209904
Title: Study on Understanding the Overall Effectiveness of Mindline.sg on Improving Mental Health Literacy, Quality of Life and Economic Outcomes
Brief Title: Economic Evaluation of Mindline.sg
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Evidence and Implementation Singapore Ltd (Other)
Collaborators: MOH Office for Healthcare Transformation (MOHT), Singapore (Unknown); National University of Singapore, Behavioural and Implementation Science Interventions (Unknown)
Responsible Party: Principal Investigator, Jean Liu, Associate Director, Centre for Evidence and Implementation Singapore Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: NUS-IRB-2025-228
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: digital mental health

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the control or intervention group.
  * Control Group: In the control group, participants will receive mental health literacy materials based on standard materials given out in Singapore (e.g., from the Health Promotion Board).
  * Intervention Group: In the intervention group, participants will be encouraged to use Mindline.sg for four weeks. The intervention includes weekly prompts to engage with different platform features,
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): In the control group, participants will receive mental health literacy materials based on standard materials given out in Singapore. At the end-of-study debrief, control group participants will be directed to the mindline.sg website so they can benefit from it.
- Intervention (Experimental): In the intervention group, participants will be encouraged to use Mindline.sg for four weeks. Each week, participants will receive a reminder to complete certain activities on the website and a quiz to measure completion of activities.
  Interventions: Behavioral: mindline.sg

INTERVENTIONS:
Behavioral: mindline.sg — mindline.sg is a polydigital mental health platform with resources, wayfinding, and peer support via a forum. The website was built by the MOH Office for Healthcare Transformation together with Ministry of Social and Family Development, National Council of Social Service and Institute of Mental health. The content was cureated by the mindline.sg team and vetted by a clinical review panel which included clinicians from IMH and Fei Yue Community Services.
  Arms: Intervention

SUMMARY:
This study aims to evaluate the effectiveness of mindline.sg, a digital mental health platform, in improving mental health literacy, emotional wellbeing, quality of life, and economic outcomes among adults in Singapore. We will conduct a randomized controlled trial (RCT) with two phases: an initial screening and a 1-month intervention. Eligible participants, identified based on mental health symptom scores, will be randomly assigned to either an intervention group using mindline.sg or a control group receiving standard mental health information.

The intervention group will receive weekly prompts to engage with key features of the platform, including psychoeducation, positive psychology tools, emotion regulation exercises, and access to digital navigation for mental health services. Participants in both groups will complete surveys at baseline, post-intervention, and two months post-intervention, measuring outcomes such as mental health symptoms, resilience, wellbeing, emotion regulation, mental health literacy, and work performance. We expect mindline.sg users to show greater improvements across mental health and quality of life indicators, increased mental health literacy, and better work productivity compared to controls. This study will provide evidence on the utility of digital mental health tools in supporting population mental wellbeing and inform future digital mental health strategies in Singapore and similar contexts.

DETAILED DESCRIPTION:
The primary hypothesis is:

- Participants in the intervention group using mindline.sg will show significantly greater improvements in mental health outcomes, quality of life, and work productivity at post-intervention (T1) and 3-month follow-up (T2), compared to the control group.

Secondary hypotheses include:

* Intervention participants will demonstrate increased resilience, better emotion regulation, and more positive attitudes and behaviors toward mental health help-seeking compared to the control group.
* Participants in the intervention group will show higher usage and engagement with digital mental health features and report higher perceived helpfulness of tools.
* The mindline.sg intervention will be cost-effective compared to the control condition, considering improvements in mental health and productivity outcomes relative to platform costs.

The study will use a randomized controllled trial design. Participants will be assigned to either: (1) A control group (receiving a mental health information pamphlet), or (2) An intervention group (using mindline.sg). Primary outcomes include mental health status, quality of life, economic and productivity measures, and user engagement metrics.

Trial participation will last 3 months. We aim to screen 5,000 adults from the general population who are aged 21 and above, have lived in Singapore for at least two years, have no psychiatric history, and are not currently receiving mental health treatment.

Participants from screening whose DASS-21 scores are mild to moderate for any one of the following sub scales will be recruited for the subsequent phase of the study.

Participants will be randomly assigned to either the control or intervention group. In the control group, participants will receive mental health literacy materials based on standard materials given out in Singapore (e.g., from the Health Promotion Board). In the intervention group, participants will be encouraged to use Mindline.sg for four weeks.

The intervention includes weekly prompts to engage with different platform features, for example:

* Week 1: Mental health literacy (Self-assessment tools and psychoeducation modules e.g. 'understand stress', 'find perspective')
* Week 2: Positive psychology and meditation exercises through Wysa AI chat (Completion of at least 4 exercises, e.g. 'Feel more control', 'be grateful', 'think motivation', 'identify your strengths', 'be kind to yourself', 'offload your worries', 'talk about your day'). Do note that Wysa's AI materials are carefully assessed for mental health appropriateness. Users can access the Wysa AI chat directly through the mindline platform without any further registration or account creation.
* Week 3: Emotion regulation exercises on mindline.sg platform (eg: tackling emotional burnout, overcoming insecurity, overcoming low mood and regaining motivation)
* Week 4: Help-seeking and personalized toolkit (explore service wayfinding tools for further mental health resources, mindline.sg live chat).

Participants will not be required to download any third party app. They are also not required to disclose any personal data during registration or use of the mindline.sg platform. Weekly activities will likely take between 10 - 30 mins, depending on the activities. Participants can exit and come back to the website later and continue their activities at their own pace. Each week, participants will receive weekly reminders via phone (e.g. messenger app) or email. This will contain infographics explaining the features.

Additionally, to ensure compliance, participants will be given a quiz at the end of each week with reimbursements for quiz completion. At the end of each week, they will also be asked to report on their use of site features (frequency and feature(s) used, and perceived helpfulness of feature), as well as their mood (three visual-analogue scales tracking: overall mood, stress, and ability to cope with challenges during the week). The quizzes will focus on participants' engagement with the platform, user experience, satisfaction, and feedback on specific features-such as what they liked or didn't like, and what worked well or didn't work. There are no "right" or "wrong" answers.

Reimbursement will be based on completeness of the quiz, not correctness-so as long as participants complete all the questions, they will be eligible.

The peer support forum feature (Let's Talk) on the mindline platform will not be part of the package as there is a separate study to evaluate it specifically.

At the end-of-study debrief, control group participants will be directed to the mindline.sg website so they too can benefit from it.

(b) Participants will also complete measures at three time-points: baseline (T0), immediately after the intervention (T1), and 2-months post-intervention. Across the three measurement timepoints, participants will be asked to complete a questionnaire to measure primary and secondary outcomes.

To provide further context, we will analyse aggregated and anonymised administrative data from the platform during the study period, including:

* Referrals: Referrals (self-reported) from mineline.sg to offline mental health services;
* Costs of mindline, including: Development and operational costs.

Please note that this project is a collaborative initiative between the Behavioural and Implementation Sciences Interventions (BISI) at YLLSoM, NUS, the Centre for Evidence and Implementation (CEI), and Ministry of Health Office for Healthcare Transformation (MOHT) formalized through a project contract signed among the three organisations. The project is supported with funding from MOHT.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 21 years or at least 18 years old if National of University student
* Have lived in Singapore for at least 2 years
* Have not received a formal diagnosis of a psychiatric disorder
* Not currently receiving any form of mental health treatment (e.g., counselling)
* Fluent in English
* Participants from screening whose DASS-21 scores are mild or moderate for any one of the sub scales.

Exclusion Criteria:

- Those who do not meet the inclusion criteria will be screened and excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Mental health symptoms by 21-item Depression, Anxiety and Stress Scale (DASS-21) | Screening, baseline, 4 weeks after baseline, 12 weeks after baseline
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest / involvement, anhedonia and inertia. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale is sensitive to levels of chronic non-specific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient. Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items. Higher scores indicate higher severity of symptoms.
Quality of Life by 6-item EQ-5D-5L scale | Baseline, 4 weeks after baseline, 12 weeks after baseline
  The 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQol Group in 2009 to improve the instrument's sensitivity and to reduce ceiling effects, as compared to the EQ-5D-3L. The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Work productivity by WHO-HPQ measure of absenteeism and presenteeism | 4 weeks after baseline, 12 weeks after baseline
  Absenteeism questions included both sickness absence and non-sickness absence. The questions asked about the number of days in the past 1 year that participants were absent due to health-related problem and non-health-related conditions separately. The questions about presenteeism asked the number of days in the past 1 year that participants had come to work while sick, felt they should take sick leave or were incapable of working with full performance.

SECONDARY OUTCOMES:
Resilience by 10-item Connor-Davidson Resilience Scale | Baseline, 4 weeks after baseline, 12 weeks after baseline
  The scale has been developed and tested as (i) a measure of degree of resilience, (ii) as a predictor of outcome to treatment with medication or psychotherapy, stress management and resilience-building; (iii) as a marker of progress during treatment; (iv) as a marker of biological (i.e. physical) changes in the brain. The scale also has promise as a method to screen people for high, intermediate or low resilience. For the CD-RISC-10, the total score ranges from 0-40.
Attitudes, knowledge and behaviours regarding mental health and help-seeking by the Mental Help Seeking Attitudes Scale (MHSAS) | Baseline, 4 weeks after baseline, 12 weeks after baseline
  The MHSAS is a 9-item instrument designed to measure respondents' overall evaluation (unfavorable vs. favorable) of their seeking help from a mental health professional if they found themselves to be dealing with a mental health concern. A higher score indicates a more positive attitude toward seeking help. The MHSAS score is a measure of help seeking attitude (Hammer, Parent, & Spiker, 2018), as it is known in the literature on professional mental health treatment seeking behavior. More precisely, the MHSAS score is a numerical quantification of the degree to which a person reports having a negative versus positive attitude toward their seeking help from a mental health professional.
Positive psychology by the Cantril Ladder and the WHO-5 Wellbeing Index | Baseline, 4 weeks after baseline, 12 weeks after baseline
  The Cantril Ladder is a question that measures life satisfaction and well-being by asking individuals to rate their current life on a scale of 0 to 10, with 10 being the best possible life and 0 being the worst.
  The WHO-5 is a self-report instrument measuring mental well-being. It consists of five statements relating to the past two weeks. Respondents rate their experiences over the past two weeks on a 6-point scale, and the total score is multiplied by 4 to create a 0-100 scale, where higher scores indicate better well-being.
Emotion regulation by DERS-18 | Baseline, 4 weeks after baseline, 12 weeks after baseline
  DERS-18 is a brief version of the Difficulties in Emotion Regulation Scale, with 18 items, and is a brief version of the original 36 item DERS. This scale measures an integrative conceptualization of emotion regulation as involving not just the modulation of emotional arousal, but also the awareness, understanding, and acceptance of emotions, and the ability to act in desired ways regardless of emotional state. The DERS-18 can be used to facilitate understanding of how emotion dysregulation is associated with psychiatric symptoms and treatment progress; it can help track changes in a client's ability to self-regulate throughout the course of treatment. Respondents rate how often they experience the statements listed (e.g., "I pay attention to how I feel") on a scale from "Almost never" to "Almost always".
Self-reported usage patterns of mindline.sg | Baseline, during intervention, 4 weeks after baseline, 12 weeks after baseline
  Frequency and features used
Cost-effectiveness of mindline.sg | Baseline, 4 weeks after baseline, 12 weeks after baseline
  The costs of the mindline.sg intervention will be cost-effective compared to the control condition, considering improvements in mental health and productivity outcomes relative to platform costs.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Liu, PhD, Principal Investigator — National University of Singapore, Yong Loo Lin School of Medicine.
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saw YE, Tan EY, Liu JS, Liu JC. Predicting Public Uptake of Digital Contact Tracing During the COVID-19 Pandemic: Results From a Nationwide Survey in Singapore. J Med Internet Res. 2021 Feb 3;23(2):e24730. doi: 10.2196/24730. PMID 33465034
- [Background] Tan EY, Wee RR, Saw YE, Heng KJ, Chin JW, Tong EM, Liu JC. Tracking Private WhatsApp Discourse About COVID-19 in Singapore: Longitudinal Infodemiology Study. J Med Internet Res. 2021 Dec 23;23(12):e34218. doi: 10.2196/34218. PMID 34881720
- [Background] Barsova T, Cheong ZG, Mak AR, Liu JC. Predicting Psychological Symptoms When Facebook's Digital Well-being Features Are Used: Cross-sectional Survey Study. JMIR Form Res. 2022 Aug 29;6(8):e39387. doi: 10.2196/39387. PMID 36036971
- [Background] Erdembileg, S., Asplund, C. L., & Liu, J. C. J. (in preparation). Engagement with Taylor Swift's music and social media content predicts mental health outcomes in youths: Cross-sectional survey study.